CLINICAL TRIAL: NCT00733980
Title: A Six-Week, Multicenter, Randomized, Double-Blind, Placebo-Controlled, Parallel-Group Study Evaluating the Efficacy, Safety, and Tolerability of GSK561679 Compared to Placebo in Female Subjects, Diagnosed With Major Depressive Disorder
Brief Title: A Study of the Effects of a New Antidepressant Treatment (GSK561679) in Females With Major Depressive Disorder
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 106139
Record Dates: First submitted 2008-08-12; First posted 2008-08-13 (Estimated); Results first posted 2017-11-17 (Actual); Last update posted 2017-11-17 (Actual); Status verified 2017-08

CONDITIONS: Depressive Disorder, Major
Keywords: Depressive Disorder, Major
MeSH Terms: conditions — Depressive Disorder, Major | interventions — NBI 77860

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- GSK561679 arm (Experimental): Double blind GSK561679
  Interventions: Drug: GSK561679
- placebo arm (Placebo Comparator): Double blind placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: GSK561679 — GSK561679
  Arms: GSK561679 arm
Other: Placebo — Placebo
  Arms: placebo arm

SUMMARY:
This six-week study will evaluate the efficacy, safety and tolerability of GSK561679 compared to placebo in female subjects with major depressive disorder

DETAILED DESCRIPTION:
This is a double-blind placebo controlled study to assess the CRF1 receptor antagonist, GSK561679, for treatment of depression in adult females diagnosed with Major Depressive Disorder (MDD). A treatment regimen of 350mg/day will be utilized to assess both efficacy and tolerability. Subjects will be randomized in equal numbers (n=75/arm) to the treatment arm and the placebo arm for a 6-week treatment period.

Efficacy will be assessed by determining the change from baseline in symptoms of MDD and anxiety utilizing the Bech Melancholia scale (Bech), Hamilton Rating Scale for Depression (HamD17), Inventory of Depressive Symptomatology-Self-Report (IDS-SR), Clinical Global Impression - Severity of Illness (CGI-S), Clinical Global Impression - Global Improvement (CGI-I), Medical Outcomes Study 12-item Sleep Module (MOS 12), Cohen Perceived Stress Test (PSS), Hamilton Anxiety Scale (HamA), and Dexamethasone Suppression Test (DST). Safety and tolerability will be assessed by determining the incidence of adverse events (AEs), vital signs, BMI, weight, clinical laboratory parameters, including ECGs, during the treatment and pre & post-treatment phases, and Discontinuation Emergent Signs and Symptoms (DESS). In addition, the incidence of suicidality will be assessed by the Columbia Suicide Severity Rating Scale (C-SSRS).

ELIGIBILITY:
Inclusion criteria:

* Female outpatients aged 25-64 years, inclusive.
* Subjects must have the ability to comprehend the consent form, and provide informed consent.
* Subject currently meets the diagnosis for MDD (without psychotic features), single episode or recurrent, as defined in the DSM-IV-TR, diagnosed with SCID-CT (Structural Clinical Interview for DSM-IV Axis I disorders - Clinical Trials Version) as assessed * by a physician with adequate training in psychiatry (e.g., Board Certification in psychiatry in the US or equivalent local qualification in other countries)
* Subject must, in the investigator's opinion based on clinical history, have met DSM IV-TR criteria for their current major depressive episode for at least 4 weeks but for no greater than 24 months.
* Subject has an IVRS HamD17 total score ≥ 23 at the Screening and Randomization Visits and the HAMD17 score is confirmed to be at least 20 by the Independent Efficacy Rater at the Screening and Randomization Visits.
* The subject is eligible to enter and participate in this study if she is not lactating and:
* Is of non-childbearing potential (i.e., physiologically incapable of becoming pregnant, including any female who is post-menopausal [defined as one year without menses]); is surgically sterile [via hysterectomy and/or removal of the ovaries] or, is of child-bearing potential, has a negative pregnancy test at both screening and baseline (prior to investigational product administration), and agrees to acceptable methods of contraception.

Exclusion Criteria

* Symptoms of the presenting illness which are better accounted for by another diagnosis*; or
* A current DSM-IV-TR Axis I diagnosis of Dementia; or
* Antisocial or Borderline Personality Disorder or other current DSM-IV-TR Axis II diagnosis that would suggest unresponsiveness to pharmacotherapy or non-compliance with the protocol; or
* A current (or within 12 months prior to the Screening visit) diagnosis of anorexia nervosa or bulimia; or
* A lifetime history of Schizophrenia, Schizoaffective Disorder, or a Bipolar Disorder.
* Subject has an unstable medical disorder or a disorder that would interfere with the action, absorption, distribution, metabolism, or excretion of GSK561679 or may pose a safety concern, or interfere with the accurate assessment of safety or efficacy.
* Subject has initiated psychotherapy within one month prior to the Screening visit, or plans to initiate psychotherapy during the trial. Subjects who present with their current MDD diagnosis despite longer-term psychotherapy (i.e., greater than three months prior to the Screening visit) and who agree to maintain the same therapy schedule during the trial may be included.
* Subject has received vagus nerve stimulation, electroconvulsive therapy, or transcranial magnetic stimulation within the six months prior to the Screening visit.
* Subject has previously failed adequate therapeutic courses of pharmacotherapy for MDD (e.g., maximum-labeled/tolerated doses for ≥ 4 weeks) from two different classes of antidepressants.
* Subject, who, in the investigator's judgement, poses a homicidal or serious suicidal risk, has had any previous suicide attempt (including aborted, interrupted or ineffective attempts) or who has ever been homicidal.
* Subject has no contact with an adult on a daily basis (i.e., subjects who are not living with at least one other adult or subjects who do not have an adult who contacts them on a daily basis). This criterion only applies to sites in Canadian sites and others where this is a local requirementa.
* Subject has a positive urine test at screening for illegal drug use and/or history of substance abuse or dependence (alcohol or drugs as defined by DSM-IV TR criteria) within the past 12 months. Subject has a blood alcohol level of ≥ 15mg/dL (0.015%) at the Screening Visit. If a subject has a positive blood alcohol or positive illegal drug results, the subject is provisionally excluded and the test cannot be repeated without prior approval of the GSK medical monitor. NOTE: Subjects must be told to avoid consumption of alcoholic beverages for at least eight hours prior to the Screening Visit. The use of alcohol by subjects participating in the study is not recommended.
* Subject has any laboratory abnormality that in the investigator's judgement is considered to be clinically significant and could potentially affect subject safety or study outcome.
* Subject has a systolic blood pressure (SBP) > 160mmHg or a diastolic blood pressure (DBP) ≥ 100 mmHg verified by repeated measurement at the Screening or Randomization visit.
* Subject is (a) currently participating in another clinical study in which the subject is or will be exposed to an investigational or non-investigational drug or device; or (b) has participated in a clinical study for an illness unrelated to depression/anxiety within the preceding month; or (c) has participated in a clinical study related to depression/anxiety within the preceding six months.
* Documented history of hepato-biliary disease including a history of, or positive laboratory results for hepatitis (hepatitis B surface antigen and/or hepatitis C antibody) at Screening, and/or clinically significant hepatic enzyme elevation 13.Subjects who are not euthyroid as evidenced by normal TSH (subjects maintained on thyroid medication must be euthyroid for a period of at least six months prior to the screen visit).
* Subject has a positive serum Human Chorionic Gonadotropin (HCG) pregnancy test at screen visit, a positive urine dipstick test at randomization, or who is lactating or planning to become pregnant within the next 13 weeks following the Screen Visit.
* Subject has clinical evidence of, or ECG results indicating any of the following at either screen or Randomization Visit unless repeat ECG shows that the parameter had returned to within normal range by the Randomisation Visit. (The ECG may be repeated to see if the parameter returns to within range):

  * QTc > 450 msec;
  * any cardiac condition or ECG evidence that the investigator feels may predispose the subject to ischemia or arrhythmia; or
  * any ECG abnormality that, in the investigator's judgment, may pose a potential safety concern.
* Subject has taken other psychoactive drugs within one week prior to the ScreeningScreening Randomization Visit
* Subject has taken systemic corticosteroids acutely within two weeks or chronically within the last 6 months of the Randomization Visit (NOTE: Topical hydrocortisone and inhaled corticosteroids are allowed).
* Subject has taken other (non-psychoactive) prescription, non-prescription, dietary, or herbal products metabolized via the cytochrome P450 3A4 pathway, or P-gp substrates with a narrow therapeutic index within 2 weeks (or 5 half-lives, whichever is longer) prior to the Randomization Visit.
* Subject has taken other (non-psychoactive) prescription, non-prescription, dietary, or herbal products that are potent inducers or inhibitors of the cytochrome P450 3A4 pathway for 2 weeks (or 5 half lives, whichever is longer) prior to the Randomization Visit.
* Subject has previously participated in an investigational trial involving GSK561679 or closely related compounds.
* Subject has a history of allergic reaction to, or significant adverse effects from excipients in the GSK561679 tablet.

Ages: 18 Years to 64 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 150 (Actual)
Dates: Start 2008-10-02 (Actual); Primary Completion 2010-06-18 (Actual); Study Completion 2010-06-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (18):
- United States (18):
  - GSK Investigational Site, Cerritos, California
  - GSK Investigational Site, San Diego, California
  - GSK Investigational Site, Torrance, California
  - GSK Investigational Site, Jacksonville, Florida
  - GSK Investigational Site, Miami, Florida
  - GSK Investigational Site, Atlanta, Georgia
  - GSK Investigational Site, Marietta, Georgia
  - GSK Investigational Site, Chicago, Illinois
  - GSK Investigational Site, Skokie, Illinois
  - GSK Investigational Site, Shreveport, Louisiana
  - GSK Investigational Site, Rockville, Maryland
  - GSK Investigational Site, Albuquerque, New Mexico
  - GSK Investigational Site, Raleigh, North Carolina
  - GSK Investigational Site, Cincinnati, Ohio
  - GSK Investigational Site, Philadelphia, Pennsylvania
  - GSK Investigational Site, Memphis, Tennessee
  - GSK Investigational Site, Brown Deer, Wisconsin
  - GSK Investigational Site, Madison, Wisconsin

REFERENCES:
- [Background] GSK has concluded that it is not feasible to publish this study in a peer-reviewed scientific journal because the nature of the study is unlikely to be of interest to a journal. GSK is providing the attached study results summary with a conclusion.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 150 female participants, with major depressive disorder (MDD), were randomized in the study. The study was conducted from 02 October 2008 to 18 June 2010 at 18 centers across the United States.
Groups:
- GSK561679: The participants in this arm received GSK561679, 350 milligram (mg) orally daily as 3x100 mg tablets plus one 50 mg tablet in evening, for 6-weeks.
- Placebo: The participants in this arm received matching placebo, and took orally as 4 placebo tablets once daily in the evening.
Period: Overall Study
Arm/Group | GSK561679 | Placebo
Started | 74 | 76
Completed | 52 | 55
Not Completed | 22 | 21
Not completed — Adverse Event | 5 | 2
Not completed — Lack of Efficacy | 0 | 1
Not completed — Protocol Violation | 2 | 1
Not completed — Protocol defined stopping criteria reach | 1 | 1
Not completed — Lost to Follow-up | 6 | 11
Not completed — Physician Decision | 2 | 3
Not completed — Withdrawal by Subject | 6 | 2

BASELINE CHARACTERISTICS:
Groups:
- GSK561679: The participants in this arm received GSK561679, 350 mg orally daily as 3x100 mg tablets plus one 50 mg tablet in evening, for 6-weeks
- Total: Total of all reporting groups
Arm/Group | GSK561679 | Placebo | Total
Number analyzed (Participants) | 74 | 76 | 150
Age, Continuous [Mean (Standard Deviation); unit: Years] | 38.8 (11.31) | 40.8 (12.17) | 39.8 (11.76)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 74 | 76 | 150
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 2 | 2
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 43 | 38 | 81
  White | 30 | 35 | 65
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change From Randomization to the End of Treatment Phase (Week 6) in the Bech Melancholia Subscale (Bech) (Items 1, 2, 7, 8, 10 and 13) From the Hamilton Rating Scale for Depression (HamD17).
Description: The Bech Melancholia Sub-scale is extracted from the HAMD-17 and is comprised of the following 6 items: Depressed Mood, Feelings of Guilt, Work and Activities, Retardation, Anxiety Psychic, and Somatic Symptoms General. The items Depressed Mood, Feelings of Guilt, Work and Activities, Retardation, Anxiety Psychic are scored on a 5-point scale from 0 to 4 except for Somatic Symptoms General which is scored on a 3-point scale from 0 to 2 where the higher scores reflecting greater severity. The Bech Melancholia Scale total score is calculated by summing the individual response scores. The highest possible score is 22 (indicative of greater severity) and the lowest possible score is 0 (indicating absence of symptoms). Change from randomization was defined as the post-baseline value minus the value at randomization. Randomization was defined as Week 0.
Time Frame: Randomization (Week 0) and Week 6
Population: Intent to Treat (ITT) population consisted of all participants who gave informed consent, were randomized, received at least one dose of double-blind medication, and had at least one post-randomization efficacy assessment available (HAM D, IDS-SR CGI, HAM A, MOS, PSS).
Measure: Least Squares Mean (Standard Error); unit: Scores on scale
Arm/Group | GSK561679 | Placebo
Number analyzed (Participants) | 72 | 74
Scores on scale | -4.3150 (0.5314) | -4.5629 (0.5101)
Statistical Analysis 1: Comparison: GSK561679 vs Placebo; Test type: Superiority or Other; p = 0.703, Mixed-Model Repeated-Measure analysis; Mean Difference (Net) = 0.2479, 80% CI [-0.5887 to 1.0846]

2. Secondary Outcome: Change From Randomization to Weeks 1, 2, and 4 in the Bech Melancholia Scale Score.
Description: The Bech Melancholia Sub-scale is extracted from the HAMD-17 and is comprised of the following 6 items: Depressed Mood, Feelings of Guilt, Work and Activities, Retardation, Anxiety Psychic, and Somatic Symptoms General. The items Depressed Mood, Feelings of Guilt, Work and Activities, Retardation, Anxiety Psychic are scored on a 5-point scale from 0 to 4 except for Somatic Symptoms General which is scored on a 3-point scale from 0 to 2 where the higher scores reflecting greater severity. The Bech Melancholia Scale total score is calculated by summing the individual response scores. The highest possible score is 22 (indicative of greater severity) and the lowest possible score is 0 (indicating absence of symptoms). Change from randomization was defined as the post-baseline value minus the value post randomization (Weeks 1, 2 and 4). Randomization was defined as Week 0.
Time Frame: Randomization (Week 0) and Week 1, 2 and 4
Population: ITT population.
Measure: Least Squares Mean (Standard Error); unit: Scores on scale
Arm/Group | GSK561679 | Placebo
Number analyzed (Participants) | 72 | 74
Scores on scale
  Week 1 | -1.6739 (0.3886) | -1.6570 (0.3540)
  Week 2 | -2.6200 (0.4436) | -3.0499 (0.4106)
  Week 4 | -3.1318 (0.4798) | -4.0731 (0.4526)
Statistical Analysis 1: Comparison: GSK561679 vs Placebo; GSK561679 Vs Placebo, Week 1; Test type: Superiority or Other; p = 0.966, Mixed Models Analysis; Mean Difference (Net) = -0.0169, 80% CI 2-sided [-0.5231 to 0.4893]
Statistical Analysis 2: Comparison: GSK561679 vs Placebo; GSK561679 Vs Placebo, Week 2; Test type: Superiority or Other; p = 0.386, Mixed Models Analysis; Mean Difference (Net) = 0.4299, 80% CI 2-sided [-0.2063 to 1.0661]
Statistical Analysis 3: Comparison: GSK561679 vs Placebo; GSK561679 Vs Placebo, Week 4; Test type: Superiority or Other; p = 0.095, Mixed Models Analysis; Mean Difference (Net) = 0.9413, 80% CI 2-sided [0.2203 to 1.6624]

3. Secondary Outcome: Change From Randomization to Weeks 1, 2, 4, and 6 in the Hamilton Anxiety Scale (HAM A)
Description: HAM A, is internationally accepted and validated measurement tool for assessment of severity of anxiety symptoms. Used to assess severity of overall anxiety in participants who met criteria for anxiety of depressive disorders and to monitor outcome of treatment. Instrument does not distinguish symptoms of specific anxiety disorder or distinguish an anxiety disorder from an anxious depression. It is clinician-administered and consists of 14 individual questions, each rated on five point scale from 0 (not present) to 4 (very severe). Total HAM A range from 0 to 56 with higher scores reflecting more severe anxiety. Change from randomization was defined as post-baseline value minus value at randomization. Randomization was defined as Week 0. Provided no more than 1 response was missing for any one visit assessment for a participant, total score was calculated adjusting for missing data as follows: Total score = (14/13)* observed total score the score was rounded to nearest integer number.
Time Frame: Randomization (Week 0) and Week 1, 2, 4 and Week 6
Population: ITT population.
Measure: Least Squares Mean (Standard Error); unit: Scores on scale
Arm/Group | GSK561679 | Placebo
Number analyzed (Participants) | 72 | 74
Scores on scale
  Week 1 | -3.4188 (0.7432) | -4.3683 (0.6649)
  Week 2 | -5.2108 (0.8347) | -5.9746 (0.7602)
  Week 4 | -5.8462 (0.9201) | -7.3825 (0.8577)
  Week 6 | -8.2330 (0.9896) | -8.8657 (0.9361)
Statistical Analysis 1: Comparison: GSK561679 vs Placebo; GSK561679 350 mg Vs Placebo, Week 1; Test type: Superiority or Other; p = 0.209, Mixed Models Analysis; Mean Difference (Net) = 0.9495, 80% CI 2-sided [-0.0185 to 1.9175]
Statistical Analysis 2: Comparison: GSK561679 vs Placebo; GSK561679 350 mg Vs Placebo, Week 2; Test type: Superiority or Other; p = 0.409, Mixed Models Analysis; Mean Difference (Net) = 0.7638, 80% CI 2-sided [-0.4243 to 1.9519]
Statistical Analysis 3: Comparison: GSK561679 vs Placebo; GSK561679 350 mg Vs Placebo, Week 4; Test type: Superiority or Other; p = 0.156, Mixed Models Analysis; Mean Difference (Net) = 1.5363, 80% CI 2-sided [0.1485 to 2.9241]
Statistical Analysis 4: Comparison: GSK561679 vs Placebo; GSK561679 350 mg Vs Placebo, Week 6; Test type: Superiority or Other; p = 0.599, Mixed Models Analysis; Mean Difference (Net) = 0.6327, 80% CI 2-sided [-0.9135 to 2.1789]

4. Secondary Outcome: Change From Randomization to Weeks 1, 2, 3, 4, and 6 in the Inventory of Depressive Symptomatology-Self- Report (IDS-SR) Total Score.
Description: The IDS-SR is self-report rating scale that assesses symptom severity of Diagnostic and Statistical Manual of Mental Disorders (DSM-IV), diagnostic criterion for major depressive disorder. The IDS-SR is a 30 item self report used to assess the severity of depressive symptoms. Each item has a 4-likert scale and each symptom item is given equivalent weightings and scored on 0 to 3 scale, with 3 representing the worst symptom. The total score of IDS-SR is calculated as a sum of each item score. The range of possible score is between 0 and 90, 0 as no symptom and 90 the worst symptom. The higher the score, the more severe the depression. Change from randomization was defined as the post-baseline value minus the value post randomization (Weeks 1, 2,3, 4 and 6). Randomization was defined as Week 0.
Time Frame: Randomization (Week 0) and Week 1, 2, 3,4 and Week 6
Population: ITT population
Measure: Least Squares Mean (Standard Error); unit: Scores on scale
Arm/Group | GSK561679 | Placebo
Number analyzed (Participants) | 72 | 74
Scores on scale
  Week 1 | -6.9509 (1.4790) | -4.9644 (1.3492)
  Week 2 | -9.9178 (1.6612) | -9.6640 (1.5354)
  Week 3 | -11.4163 (1.7251) | -11.0921 (1.6115)
  Week 4 | -12.3463 (1.9146) | -13.1571 (1.8066)
  Week 6 | -15.5045 (2.0467) | -14.8772 (1.9522)
Statistical Analysis 1: Comparison: GSK561679 vs Placebo; GSK561679 350 mg Vs Placebo, Week 1; Test type: Superiority or Other; p = 0.181, Mixed Models Analysis; Mean Difference (Net) = -1.9866, 80% CI 2-sided [-3.8876 to -0.0856]
Statistical Analysis 2: Comparison: GSK561679 vs Placebo; GSK561679 350 mg Vs Placebo, Week 2; Test type: Superiority or Other; p = 0.889, Mixed Models Analysis; Mean Difference (Net) = -0.2538, 80% CI 2-sided [-2.5922 to 2.0846]
Statistical Analysis 3: Comparison: GSK561679 vs Placebo; GSK561679 350 mg Vs Placebo, Week 3; Test type: Superiority or Other; p = 0.867, Mixed Models Analysis; Mean Difference (Net) = -0.3242, 80% CI 2-sided [-2.8165 to 2.1681]
Statistical Analysis 4: Comparison: GSK561679 vs Placebo; GSK561679 350 mg Vs Placebo, Week 4; Test type: Superiority or Other; p = 0.721, Mixed Models Analysis; Mean Difference (Net) = 0.8107, 80% CI 2-sided [-2.1036 to 3.7251]
Statistical Analysis 5: Comparison: GSK561679 vs Placebo; GSK561679 350 mg Vs Placebo, Week 6; Test type: Superiority or Other; p = 0.801, Mixed Models Analysis; Mean Difference (Net) = -0.6273, 80% CI 2-sided [-3.8337 to 2.5791]

5. Secondary Outcome: Change From Randomization to Weeks 1, 2, 4, and 6 in the Hamilton Rating Scale for Depression (HAMD-17)
Description: The HAMD-17 scale is a subset of HAMD-28. It is a standard used to measure depression severity. The HAMD-17 score ranges from 0 to 52; a score of 0-7 is generally accepted to be within the normal range (or in clinical remission), while a score of 20 or higher indicates at least moderate severity; a reduction of 50% or more in total score from Baseline indicates clinical response. Thus a higher score was indicative of more severity. Change from randomization was defined as the post-baseline value minus the value at randomization. Randomization was defined as Week 0.
Time Frame: Randomization (Week 0) and Week 1, 2, 4 and Week 6
Population: ITT population.
Measure: Least Squares Mean (Standard Error); unit: Scores on scale
Arm/Group | GSK561679 | Placebo
Number analyzed (Participants) | 72 | 74
Scores on scale
  Week 1 | -3.6342 (0.6816) | -4.2782 (0.6198)
  Week 2 | -5.1998 (0.8009) | -6.2523 (0.7425)
  Week 4 | -6.5337 (0.8734) | -8.1810 (0.8262)
  Week 6 | -8.2503 (0.9770) | -8.9786 (0.9376)
Statistical Analysis 1: Comparison: GSK561679 vs Placebo; GSK561679 350 mg Vs Placebo, Week 1; Test type: Superiority or Other; p = 0.355, Mixed Models Analysis; Mean Difference (Net) = 0.6440, 80% CI 2-sided [-0.2498 to 1.5378]
Statistical Analysis 2: Comparison: GSK561679 vs Placebo; GSK561679 350 mg Vs Placebo, Week 2; Test type: Superiority or Other; p = 0.249, Mixed Models Analysis; Mean Difference (Net) = 1.0524, 80% CI 2-sided [-0.1194 to 2.2243]
Statistical Analysis 3: Comparison: GSK561679 vs Placebo; GSK561679 350 mg Vs Placebo, Week 4; Test type: Superiority or Other; p = 0.116, Mixed Models Analysis; Mean Difference (Net) = 1.6473, 80% CI 2-sided [0.3078 to 2.9868]
Statistical Analysis 4: Comparison: GSK561679 vs Placebo; GSK561679 350 mg Vs Placebo, Week 6; Test type: Superiority or Other; p = 0.550, Mixed Models Analysis; Mean Difference (Net) = 0.7283, 80% CI 2-sided [-0.8353 to 2.2920]

6. Secondary Outcome: Percentage HAMD-17 Responders at Weeks 1, 2, 4, and 6.
Description: HAMD-17 Responders were defined as the participants with a > or = 50% reduction from randomization in their HAMD-17 total score at Weeks 1, 2, 4, and 6. The HAMD-17 scale is a subset of HAMD-28. It is a standard used to measure depression severity. The HAMD-17 score ranged from 0 to 52; a score of 0-7 is generally accepted to be within the normal range (or in clinical remission), while a score of 20 or higher indicated at least moderate severity; a reduction of 50% or more in total score from Baseline indicates clinical response. Thus a higher score was indicative of more severity.
Time Frame: Weeks 1, 2, 4, and 6.
Population: ITT population. Only those participants available at the specified time points were analyzed.
Measure: Number; unit: Percentage of participants
Arm/Group | GSK561679 | Placebo
Number analyzed (Participants) | 71 | 74
Percentage of participants
  Week 1 | 3 | 4
  Week 2 | 7 | 15
  Week 4 | 17 | 24
  Week 6 | 27 | 28

7. Secondary Outcome: Time to Maintained Antidepressant Response at the End of Treatment Phase (Week 6)
Description: The time to maintained antidepressant response at the end of treatment phase (week 6), as the participants with a > or = to 50 % reduction from randomization in their HAMD-17 total score, sustained until the end of the Treatment Phase [Week 6]). This OM "time to maintained antidepressant response" was not evaluated due to lower number of participants in the GSK561679 group as compared to placebo
Time Frame: Week 6
Population: Endpoint not evaluated.
Arm/Group | GSK561679 | Placebo
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Change From Randomization in the Clinical Global Impression - Severity of Illness (CGI-S) Score at Weeks 1, 2, 4, and 6.
Description: The CGI is a widely accepted measure of illness severity and clinical improvement in a variety of psychiatric disorders. The CGI is psychiatrist rated, and is based on all information available at the time of the rating. Both the CGI-I and CGI-S items are rated on a 1 to 7 point scale. Scores on the CGI-I range from 1 (very much improved) to 7 (very much worse). Scores, on the CGI-S, range from 1 (normal, not ill at all) to 7 (amongst the most extremely ill). Change from randomization was defined as the post-baseline value minus the value at randomization. Randomization was defined as Week 0.
Time Frame: Randomization (Week 0) and Weeks 1, 2, 4, and 6.
Population: ITT population
Measure: Least Squares Mean (Standard Error); unit: Scores on scale
Arm/Group | GSK561679 | Placebo
Number analyzed (Participants) | 72 | 74
Scores on scale
  Week 1 | -0.2800 (0.0859) | -0.2632 (0.0783)
  Week 2 | -0.4013 (0.1026) | -0.4677 (0.0957)
  Week 4 | -0.5866 (0.1222) | -0.9557 (0.1169)
  Week 6 | -0.8353 (0.1384) | -1.1103 (0.1348)

9. Secondary Outcome: Percentage of Clinical Global Impression - Global Improvement (CGI-I) Responders at Weeks 1, 2, 4, and 6.
Description: The CGI is a widely accepted measure of illness severity and clinical improvement in a variety of psychiatric disorders. The CGI is psychiatrist rated, and is based on all information available at the time of the rating. The CGI -responders, are defined as participants with a score of 1 (very much improved) or 2 (much improved) in the CGI-I).
Time Frame: Weeks 1, 2, 4, and 6.
Measure: Number; unit: perecntage of participants
Arm/Group | GSK561679 | Placebo
Number analyzed (Participants) | 72 | 74
perecntage of participants
  Week 1 | 3 | 5
  Week 2 | 11 | 16
  Week 4 | 25 | 32
  Week 6 | 33 | 36
Statistical Analysis 1: Comparison: GSK561679 vs Placebo; GSK561679 350 mg Vs Placebo, Week 2; Test type: Superiority or Other; p = 0.3588, Logistic Model; Odds Ratio (OR) = 0.6359, 80% CI 2-sided [0.3378 to 1.1968]
Statistical Analysis 2: Comparison: GSK561679 vs Placebo; GSK561679 350 mg Vs Placebo, Week 4; Test type: Superiority or Other; p = 0.4088, Logistic Model; Odds Ratio (OR) = 0.7347, 80% CI 2-sided [0.4554 to 1.1853]
Statistical Analysis 3: Comparison: GSK561679 vs Placebo; GSK561679 350 mg Vs Placebo, Week 6/ Early withdrawal; Test type: Superiority or Other; p = 0.8156, Logistic Model; Logistic Model = 0.9211, 80% CI 2-sided [0.5863 to 1.4471]

10. Secondary Outcome: Change From Randomization in the Medical Outcomes Study 12-item Sleep Module (MOS 12) at Week 6
Description: The MOS-12 Sleep Scale is a 12-item questionnaire which measures specific aspects of sleep in participants that may have varying co-morbidities, as a result, is appropriate for a medically diverse participant population. It consist of following items: initiation (2 items), maintenance (2 items), respiratory problems (2 items), quantity (1 item), perceived adequacy (2 items), and somnolence (3 items). All items were given equivalent weightage from 1 to 6. Each index summarizes information across most or all sleep dimensions. The total score is transformed linearly to a common metric with a possible range of 0-100 and is averaged across items in the same scale. The higher score indicates a greater degree of the attribute implied by the scale name. Change from randomization was calculated by randomization value minus the value at Week 6. Randomization was defined as Week 0.
Time Frame: Randomization (Week 0) and Week 6
Population: ITT population.
Measure: Least Squares Mean (Standard Error); unit: Scores on scale
Arm/Group | GSK561679 | Placebo
Number analyzed (Participants) | 72 | 74
Scores on scale | -16.2738 (3.7112) | -19.7203 (3.4794)
Statistical Analysis 1: Comparison: GSK561679 vs Placebo; Test type: Superiority or Other; p = 0.361, ANCOVA; Mean Difference (Net) = 3.4466, 80% CI 2-sided [-1.3986 to 8.2917]

11. Secondary Outcome: Change From Randomization in the Cohen Perceived Stress Scale (PSS) at Week 6.
Description: The PSS is most widely used psychological instrument for measuring the perception of stress. It is a 10-item questionnaire that measures an individual's subjective evaluation the stressfulness of situations in their life in past month (how unpredictable, uncontrollable, and overloaded respondents find their lives). Individual items were rated on a scale of 0-4, where 0(never) to 4 (very often) that best describes how often they have had the feelings or thoughts described in the last month for each question. The total scores can range from 0-40, where 0 score indicated no stress and a higher score indicated more stress. Change from randomization was defined as the post-baseline value minus the value at randomization. Randomization was defined as Week 0. Thus a negative change from randomization indicated improvement.
Time Frame: Randomization (Week 0) and Week 6.
Population: ITT population.
Measure: Least Squares Mean (Standard Error); unit: Scores on scale
Arm/Group | GSK561679 | Placebo
Number analyzed (Participants) | 72 | 74
Scores on scale | -5.6529 (1.3431) | -5.7696 (1.2624)
Statistical Analysis 1: Comparison: GSK561679 vs Placebo; Test type: Superiority or Other; p = 0.932, ANCOVA; Mean Difference (Net) = 0.1167, 80% CI 2-sided [-1.6387 to 1.8722]

12. Secondary Outcome: Number of Participants With Adverse Events (AE) and Serious Adverse Events (SAE)
Description: An AE was any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a medicinal (investigational) product, whether or not considered related to the medicinal (investigational) product. For marketed medicinal products, this also includes failure to produce expected benefits (i.e. lack of efficacy), abuse or misuse. SAE was any experience that: resulted in death, was life-threatening, required in-patient hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity, was a congenital anomaly/birth defect or was medically significant.
Time Frame: Up to 28-day FU (18 months)
Population: All subject population.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK561679 | Placebo
Number analyzed (Participants) | 74 | 76
Participants
  Any AE | 55 | 58
  Any SAE | 0 | 1

13. Secondary Outcome: Number of Participants With Vital Sign of Potential Clinical Importance (PCI)
Description: Vital sign measurements included height (screening only), systolic blood pressure(SBP) and diastolic blood pressure (DBP) and heart rate (HR). Sitting vital signs were measured at all clinic visits. Standing vital signs were measured at screening, Week 3 and at any other times as clinically indicated. Only the PCI values for SBP, DBP and HR were reported.
Time Frame: Up to Week 10
Population: All subject population.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK561679 | Placebo
Number analyzed (Participants) | 74 | 76
Participants
  SBP, High | 1 | 2
  SBP, Low | 2 | 3
  DBP, HIgh | 7 | 4
  DBP, Low | 1 | 0
  HR, High | 1 | 2

14. Secondary Outcome: Number of Participants With Abnormal Urinalysis Data
Description: Urinalysis included analysis for urine bilirubin, urine occult blood, urine glucose, urine ketones, urine nitrite, urine proteins and urine Leukocyte Esterase test (LET) via dipstick analysis. The number of participants with abnormal urinalysis data were reported. In the dipstick test the levels for urine bilirubin, urine occult blood, urine glucose, urine ketones, urine nitrite, urine proteins and urine LET with results of trace, negative, positive,1+=slightly positive, 2+=positive, 3+=high positive were reported.
Time Frame: Randomization (Week 0), Week 3, Week 6/ Early withdrawal (EW) and 28 Day follow-up (FU)
Population: All subject population.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK561679 | Placebo
Number analyzed (Participants) | 74 | 76
Participants
  Urine Bilirubin, Randomized, negative: number analyzed (Participants) | 74 | 74
  Urine Bilirubin, Randomized, negative | 74 | 74
  Urine Occult Blood, Randomized, 1+: number analyzed (Participants) | 74 | 74
  Urine Occult Blood, Randomized, 1+ | 3 | 3
  Urine Occult Blood, Randomized, 2+: number analyzed (Participants) | 74 | 74
  Urine Occult Blood, Randomized, 2+ | 6 | 2
  Urine Occult Blood, Randomized, 3+: number analyzed (Participants) | 74 | 74
  Urine Occult Blood, Randomized, 3+ | 2 | 2
  Urine Occult Blood, Randomized, negative: number analyzed (Participants) | 74 | 74
  Urine Occult Blood, Randomized, negative | 58 | 63
  Urine Occult Blood, Randomized, trace: number analyzed (Participants) | 74 | 74
  Urine Occult Blood, Randomized, trace | 5 | 4
  Urine Glucose, Randomized, 2+: number analyzed (Participants) | 74 | 74
  Urine Glucose, Randomized, 2+ | 1 | 1
  Urine Glucose, Randomized, 3+: number analyzed (Participants) | 74 | 74
  Urine Glucose, Randomized, 3+ | 0 | 1
  Urine Glucose, Randomized, negative: number analyzed (Participants) | 74 | 74
  Urine Glucose, Randomized, negative | 73 | 71
  Urine Glucose, Randomized, trace: number analyzed (Participants) | 74 | 74
  Urine Glucose, Randomized, trace | 0 | 1
  Urine Ketones, Randomized, negative: number analyzed (Participants) | 74 | 74
  Urine Ketones, Randomized, negative | 73 | 71
  Urine Ketones, Randomized, trace: number analyzed (Participants) | 74 | 74
  Urine Ketones, Randomized, trace | 1 | 3
  Urine Nitrite, Randomized, negative: number analyzed (Participants) | 74 | 74
  Urine Nitrite, Randomized, negative | 73 | 71
  Urine Nitrite, Randomized, positive: number analyzed (Participants) | 74 | 74
  Urine Nitrite, Randomized, positive | 1 | 3
  Urine Protein, Randomized, 1+: number analyzed (Participants) | 74 | 74
  Urine Protein, Randomized, 1+ | 3 | 4
  Urine Protein, Randomized, negative: number analyzed (Participants) | 74 | 74
  Urine Protein, Randomized, negative | 64 | 61
  Urine Protein, Randomized, trace: number analyzed (Participants) | 74 | 74
  Urine Protein, Randomized, trace | 7 | 9
  Urine LET for WBC, Randomized, 1+: number analyzed (Participants) | 74 | 74
  Urine LET for WBC, Randomized, 1+ | 5 | 3
  Urine LET for WBC, Randomized, 2+: number analyzed (Participants) | 74 | 74
  Urine LET for WBC, Randomized, 2+ | 4 | 7
  Urine LET for WBC, Randomized, 3+: number analyzed (Participants) | 74 | 74
  Urine LET for WBC, Randomized, 3+ | 1 | 1
  Urine LET for WBC, Randomized, negative: number analyzed (Participants) | 74 | 74
  Urine LET for WBC, Randomized, negative | 60 | 59
  Urine LET for WBC, Randomized, trace: number analyzed (Participants) | 74 | 74
  Urine LET for WBC, Randomized, trace | 4 | 4
  Urine bilirubin, Week 3, negative: number analyzed (Participants) | 60 | 63
  Urine bilirubin, Week 3, negative | 60 | 63
  Urine Occult Blood, Week 3, 1+: number analyzed (Participants) | 60 | 63
  Urine Occult Blood, Week 3, 1+ | 3 | 3
  Urine Occult Blood, Week 3, 2+: number analyzed (Participants) | 60 | 63
  Urine Occult Blood, Week 3, 2+ | 2 | 1
  Urine Occult Blood, Week 3, 3+: number analyzed (Participants) | 60 | 63
  Urine Occult Blood, Week 3, 3+ | 1 | 0
  Urine Occult Blood, Week 3, negative: number analyzed (Participants) | 60 | 63
  Urine Occult Blood, Week 3, negative | 53 | 57
  Urine Occult Blood, Week 3, trace: number analyzed (Participants) | 60 | 63
  Urine Occult Blood, Week 3, trace | 1 | 2
  Urine Glucose, Negative: number analyzed (Participants) | 60 | 63
  Urine Glucose, Negative | 60 | 63
  Urine Ketones, Week 3, 1+: number analyzed (Participants) | 60 | 63
  Urine Ketones, Week 3, 1+ | 0 | 1
  Urine Ketones, Week 3, negative: number analyzed (Participants) | 60 | 63
  Urine Ketones, Week 3, negative | 55 | 61
  Urine Ketones, Week 3, trace: number analyzed (Participants) | 60 | 63
  Urine Ketones, Week 3, trace | 5 | 1
  Urine nitrite, Week 3, negative: number analyzed (Participants) | 60 | 63
  Urine nitrite, Week 3, negative | 60 | 60
  Urine nitrite, Week 3, positive: number analyzed (Participants) | 60 | 63
  Urine nitrite, Week 3, positive | 0 | 3
  Urine Protein, Week 3, 1+: number analyzed (Participants) | 60 | 63
  Urine Protein, Week 3, 1+ | 4 | 1
  Urine Protein, Week 3, negative: number analyzed (Participants) | 60 | 63
  Urine Protein, Week 3, negative | 46 | 53
  Urine Protein, Week 3, positive: number analyzed (Participants) | 60 | 63
  Urine Protein, Week 3, positive | 10 | 9
  Urine LET for WBC, Week 3, 1+: number analyzed (Participants) | 60 | 63
  Urine LET for WBC, Week 3, 1+ | 3 | 5
  Urine LET for WBC, Week 3, 2+: number analyzed (Participants) | 60 | 63
  Urine LET for WBC, Week 3, 2+ | 3 | 2
  Urine LET for WBC, Week 3, 3+: number analyzed (Participants) | 60 | 63
  Urine LET for WBC, Week 3, 3+ | 1 | 1
  Urine LET for WBC, Week 3, negative: number analyzed (Participants) | 60 | 63
  Urine LET for WBC, Week 3, negative | 51 | 48
  Urine LET for WBC, Week 3, trace: number analyzed (Participants) | 60 | 63
  Urine LET for WBC, Week 3, trace | 2 | 7
  Urine Bilirubin, Week 6/EW, negative: number analyzed (Participants) | 69 | 65
  Urine Bilirubin, Week 6/EW, negative | 69 | 65
  Urine Occult Blood, Week 6/EW, 1+: number analyzed (Participants) | 69 | 65
  Urine Occult Blood, Week 6/EW, 1+ | 2 | 2
  Urine Occult Blood, Week 6/EW, 2+: number analyzed (Participants) | 69 | 65
  Urine Occult Blood, Week 6/EW, 2+ | 1 | 3
  Urine Occult Blood, Week 6/EW, 3+: number analyzed (Participants) | 69 | 65
  Urine Occult Blood, Week 6/EW, 3+ | 9 | 2
  Urine Occult Blood, Week 6/EW, negative: number analyzed (Participants) | 69 | 65
  Urine Occult Blood, Week 6/EW, negative | 54 | 56
  Urine Occult Blood, Week 6/EW, trace: number analyzed (Participants) | 69 | 65
  Urine Occult Blood, Week 6/EW, trace | 3 | 2
  Urine Glucose, Week 6/EW, negative: number analyzed (Participants) | 69 | 65
  Urine Glucose, Week 6/EW, negative | 69 | 65
  Urine ketone, Week 6/EW, negative: number analyzed (Participants) | 69 | 65
  Urine ketone, Week 6/EW, negative | 64 | 63
  Urine ketone, Week 6/EW, trace: number analyzed (Participants) | 69 | 65
  Urine ketone, Week 6/EW, trace | 5 | 2
  Urine Nitrite, Week 6/EW, negative: number analyzed (Participants) | 69 | 65
  Urine Nitrite, Week 6/EW, negative | 68 | 62
  Urine Nitrite, Week 6/EW, positive: number analyzed (Participants) | 69 | 65
  Urine Nitrite, Week 6/EW, positive | 1 | 3
  Urine protein, Week 6/EW, 1+: number analyzed (Participants) | 69 | 65
  Urine protein, Week 6/EW, 1+ | 7 | 4
  Urine protein, Week 6/EW, 2+: number analyzed (Participants) | 69 | 65
  Urine protein, Week 6/EW, 2+ | 2 | 1
  Urine protein, Week 6/EW, negative: number analyzed (Participants) | 69 | 65
  Urine protein, Week 6/EW, negative | 52 | 55
  Urine protein, Week 6/EW, trace: number analyzed (Participants) | 69 | 65
  Urine protein, Week 6/EW, trace | 8 | 5
  Urine LET for WBC , Week 6/EW, 1+: number analyzed (Participants) | 69 | 65
  Urine LET for WBC , Week 6/EW, 1+ | 6 | 4
  Urine LET for WBC, Week 6/EW, 2+ | 1 | 4
  Urine LET for WBC, Week 6/EW, 3+ | 4 | 2
  Urine LET for WBC, Week 6/EW, negative | 51 | 53
  Urine LET for WBC, Week 6/EW, trace | 7 | 2
  Urine Bilirubin, 28-day FU, negative: number analyzed (Participants) | 18 | 17
  Urine Bilirubin, 28-day FU, negative | 18 | 17
  Urine Occult Blood, 28-day FU, 1+: number analyzed (Participants) | 18 | 17
  Urine Occult Blood, 28-day FU, 1+ | 1 | 2
  Urine Occult Blood, 28-day FU, 2+: number analyzed (Participants) | 18 | 17
  Urine Occult Blood, 28-day FU, 2+ | 1 | 1
  Urine Occult Blood, 28-day FU, 3+: number analyzed (Participants) | 18 | 17
  Urine Occult Blood, 28-day FU, 3+ | 2 | 0
  Urine Occult Blood, 28-day FU, negative: number analyzed (Participants) | 18 | 17
  Urine Occult Blood, 28-day FU, negative | 13 | 13
  Urine Occult Blood, 28-day FU, trace: number analyzed (Participants) | 18 | 17
  Urine Occult Blood, 28-day FU, trace | 1 | 1
  Urine Glucose, 28-day FU, negative: number analyzed (Participants) | 18 | 17
  Urine Glucose, 28-day FU, negative | 18 | 17
  Urine Ketones, 28-day FU, 1+: number analyzed (Participants) | 18 | 17
  Urine Ketones, 28-day FU, 1+ | 0 | 1
  Urine Ketones, 28-day FU, negative: number analyzed (Participants) | 18 | 17
  Urine Ketones, 28-day FU, negative | 18 | 16
  Urine Nitrite, 28-day FU, negative: number analyzed (Participants) | 18 | 17
  Urine Nitrite, 28-day FU, negative | 18 | 17
  Urine Protein, 28-day FU, 1+: number analyzed (Participants) | 18 | 17
  Urine Protein, 28-day FU, 1+ | 2 | 1
  Urine Protein, 28-day FU, 2+: number analyzed (Participants) | 18 | 17
  Urine Protein, 28-day FU, 2+ | 0 | 1
  Urine Protein, 28-day FU, negative: number analyzed (Participants) | 18 | 17
  Urine Protein, 28-day FU, negative | 13 | 14
  Urine Protein, 28-day FU, trace: number analyzed (Participants) | 18 | 17
  Urine Protein, 28-day FU, trace | 3 | 1
  Urine LET for WBC, 28-day FU, 1+: number analyzed (Participants) | 18 | 17
  Urine LET for WBC, 28-day FU, 1+ | 2 | 0
  Urine LET for WBC, 28-day FU, 2+: number analyzed (Participants) | 18 | 17
  Urine LET for WBC, 28-day FU, 2+ | 1 | 2
  Urine LET for WBC, 28-day FU, 3+: number analyzed (Participants) | 18 | 17
  Urine LET for WBC, 28-day FU, 3+ | 1 | 1
  Urine LET for WBC, 28-day FU, negative: number analyzed (Participants) | 18 | 17
  Urine LET for WBC, 28-day FU, negative | 12 | 13
  Urine LET for WBC, 28-day FU, trace: number analyzed (Participants) | 18 | 17
  Urine LET for WBC, 28-day FU, trace | 2 | 1

15. Secondary Outcome: Number of Participants With Abnormal Electrocardiograph (ECG) Values
Description: The 12-lead ECG, were obtained at each time-point during the study using an ECG machine. The number of participants with ECG abnormal values were reported.
Time Frame: Randomization (Week 0), Week 4, Week 6 and 28 Day follow-up
Population: All subject population. Only those participants available at the specified time points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK561679 | Placebo
Number analyzed (Participants) | 74 | 76
Participants
  Abnormal, Randomization | 6 | 11
  Abnormal, Week 4: number analyzed (Participants) | 55 | 58
  Abnormal, Week 4 | 7 | 10
  Abnormal, Week 6/EW: number analyzed (Participants) | 70 | 65
  Abnormal, Week 6/EW | 6 | 13
  Abnormal, 28-day FU: number analyzed (Participants) | 11 | 17
  Abnormal, 28-day FU | 1 | 5

16. Secondary Outcome: Number of Participants With Abnormal Hematology Values of PCI-Platelet
Description: Number of participants with abnormal Hematology values of PCI were reported. The abnormal values were reported only for platelet, diagnosed at Week 6 or Early withdrawal visit.
Time Frame: Upto 28-day FU
Population: All Subject population
Measure: Count of Participants; unit: Participants
Arm/Group | GSK561679 | Placebo
Number analyzed (Participants) | 66 | 63
Participants | 0 | 1

17. Secondary Outcome: Number of Participants With Clinical Chemistry Laboratory Data Outside Reference Range
Description: The number of participants with clinical chemistry values outside the clinical importance range (CIR) were reported. The values for chemistry parameters outside CRI were reported for Alanine amino transferase (ALT), Aspartate amino transferase, total bilirubin, calcium, Creatine Kinase, carbon dioxide (CO^2) content/bicarbonate (BC), glucose and potassium were reported.
Time Frame: Upto Week 10
Population: All subject population.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK561679 | Placebo
Number analyzed (Participants) | 74 | 76
Participants
  ALT, Week 4, CIR, high: number analyzed (Participants) | 65 | 64
  ALT, Week 4, CIR, high | 0 | 1
  AST, Week 4, CIR, high: number analyzed (Participants) | 65 | 64
  AST, Week 4, CIR, high | 0 | 1
  Total bilirubin, Randomization, CIR, high | 0 | 1
  Total bilirubin, Week 2, CIR, high | 0 | 1
  Total bilirubin, Week 6/EW, CIR, high | 0 | 1
  Calcium, 28-day FU,CIR, low: number analyzed (Participants) | 27 | 22
  Calcium, 28-day FU,CIR, low | 0 | 1
  Creatine Kinase , Randomization, CIR,high: number analyzed (Participants) | 74 | 75
  Creatine Kinase , Randomization, CIR,high | 1 | 1
  Creatine Kinase, Week 1, CIR, high: number analyzed (Participants) | 69 | 69
  Creatine Kinase, Week 1, CIR, high | 0 | 1
  Creatine Kinase, Week 2, CIR, high: number analyzed (Participants) | 68 | 70
  Creatine Kinase, Week 2, CIR, high | 2 | 1
  Creatine Kinase, 28-day FU, CIR, high: number analyzed (Participants) | 28 | 22
  Creatine Kinase, 28-day FU, CIR, high | 1 | 0
  CO^2 content/BC, 28-day FU,CIR, low: number analyzed (Participants) | 27 | 22
  CO^2 content/BC, 28-day FU,CIR, low | 0 | 1
  Glucose, Randomization, CIR, high | 0 | 1
  Glucose, Week 6/EW, CIR, low: number analyzed (Participants) | 69 | 66
  Glucose, Week 6/EW, CIR, low | 0 | 1
  Glucose, 28-day FU,CIR, low: number analyzed (Participants) | 28 | 22
  Glucose, 28-day FU,CIR, low | 1 | 0
  Potassium, Randomization, CIR, low | 1 | 0
  Potassium, 28-day FU, CIR, high | 0 | 1

18. Secondary Outcome: Number of Participants With Hormonal Data of PCI
Description: The number of participants with hormone values outside the CRI were reported. The hormone data was analyzed for parameters like Cortisol total, Dehydroepiandrosterone, Thyroxine, free, and thyroid stimulating hormone (TSH) .
Time Frame: up to Week 10
Population: All subject population.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK561679 | Placebo
Number analyzed (Participants) | 74 | 76
Participants
  Cortisol, total, Randomization, CIR, low: number analyzed (Participants) | 73 | 76
  Cortisol, total, Randomization, CIR, low | 1 | 4
  Cortisol, total, Week 2, CIR, low: number analyzed (Participants) | 68 | 71
  Cortisol, total, Week 2, CIR, low | 0 | 1
  Cortisol, total, Week 4, CIR, low: number analyzed (Participants) | 65 | 65
  Cortisol, total, Week 4, CIR, low | 1 | 1
  Cortisol, total, Week 6/EW, CIR, low: number analyzed (Participants) | 69 | 66
  Cortisol, total, Week 6/EW, CIR, low | 1 | 0
  Dehydroepiandrosterone, Randomization, CIR, high | 0 | 2
  Dehydroepiandrosterone, Randomization, CIR, low | 3 | 5
  Dehydroepiandrosterone, Week 2, CIR, high: number analyzed (Participants) | 68 | 71
  Dehydroepiandrosterone, Week 2, CIR, high | 1 | 0
  Dehydroepiandrosterone, Week 2, CIR, low: number analyzed (Participants) | 68 | 71
  Dehydroepiandrosterone, Week 2, CIR, low | 3 | 4
  Dehydroepiandrosterone , Week 4, CIR, low: number analyzed (Participants) | 65 | 64
  Dehydroepiandrosterone , Week 4, CIR, low | 4 | 8
  Dehydroepiandrosterone, Week 6/EW, CIR, low: number analyzed (Participants) | 69 | 66
  Dehydroepiandrosterone, Week 6/EW, CIR, low | 5 | 6
  Dehydroepiandrosterone, 28-day FU,CIR, low: number analyzed (Participants) | 17 | 13
  Dehydroepiandrosterone, 28-day FU,CIR, low | 1 | 0
  Thyroxine, free, Week 6/EW, CIR, low: number analyzed (Participants) | 69 | 66
  Thyroxine, free, Week 6/EW, CIR, low | 1 | 2
  Thyroxine, free, 28-day FU,CIR, low: number analyzed (Participants) | 27 | 20
  Thyroxine, free, 28-day FU,CIR, low | 1 | 2
  TSH, Week 6/EW, CIR, high: number analyzed (Participants) | 69 | 66
  TSH, Week 6/EW, CIR, high | 0 | 1
  TSH, Week 6/EW, CIR, low: number analyzed (Participants) | 69 | 66
  TSH, Week 6/EW, CIR, low | 0 | 3
  TSH, 28-day FU, CIR, high: number analyzed (Participants) | 27 | 20
  TSH, 28-day FU, CIR, high | 1 | 1

19. Secondary Outcome: Discontinuation-Emergent Signs and Symptoms
Description: The discontinuation signs and symptoms scale consisted of 43 signs and symptoms, scored as 'new symptom (NS)', 'old symptom (OS) but worse', 'OS but improved' or ' symptom not present/old symptom but unchanged'. The total number of new signs and symptoms, old symptoms but worse, and old symptoms but improved was calculated for each participant. The number of participants with Discontinuation-Emergent Signs and Symptoms were reported. The visits were at Week 6 Visit, 7-D FU and 28-D FU visit.
Time Frame: At Week 6, 7-day (D) FU and 28-D FU
Population: All subject population.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK561679 | Placebo
Number analyzed (Participants) | 74 | 76
Participants
  Anxiety , Week 6/EW, NS | 1 | 1
  Anxiety , Week 6/EW, OS but worse | 7 | 4
  Anxiety , Week 6/EW, OS but improved | 13 | 14
  Anxiety , Week 6/EW, OS but unchanged/absent | 48 | 47
  Anxiety , 7-D FU, NS | 3 | 2
  Anxiety , 7-D FU, OS but worse | 4 | 4
  Anxiety , 7-D FU, OS but improved | 11 | 11
  Anxiety , 7-D FU, OS but unchanged/absent | 47 | 45
  Anxiety , 28-D FU, NS | 3 | 3
  Anxiety , 28-D FU, OS but worse | 9 | 6
  Anxiety , 28-D FU, OS but improved | 11 | 13
  Anxiety , 28-D FU, OS but unchanged/absent | 35 | 37
  Feeling high, Week 6/EW, NS | 0 | 2
  Feeling high, Week 6/EW, OS but worse | 1 | 1
  Feeling high, Week 6/EW, OS but improved | 5 | 6
  Feeling high, Week 6/EW, OS but unchanged/absent | 63 | 56
  Feeling high , Week 6/EW, Missing | 0 | 1
  Feeling high, 7-D FU, NS | 3 | 1
  Feeling high, 7-D FU, OS but worse | 0 | 2
  Feeling high, 7-D FU, OS but improved | 5 | 4
  Feeling high, 7-D FU, OS but unchanged/absent | 57 | 55
  Feeling high , 28-D FU, NS | 2 | 0
  Feeling high , 28-D FU, OS but worse | 2 | 1
  Feeling high , 28-D FU, OS but improved | 6 | 6
  Feeling high , 28-D FU, OS but unchanged/absent | 48 | 52
  Irritability, Week 6/EW, NS | 1 | 2
  Irritability, Week 6/EW, OS but worse | 8 | 7
  Irritability, Week 6/EW, OS but improved | 17 | 18
  Irritability, Week 6/EW, OS but unchanged/absent | 43 | 39
  Irritability, 7-D FU, NS | 1 | 2
  Irritability, 7-D FU, OS but worse | 7 | 9
  Irritability, 7-D FU, OS but improved | 12 | 13
  Irritability, 7-D FU, OS unchanged/absent | 45 | 38
  Irritability, 28-D FU, NS | 2 | 1
  Irritability, 28-D FU, OS but worse | 8 | 10
  Irritability, 28-D FU, OS but improved | 11 | 10
  Irritability, 28-D FU, OS but unchanged/absent | 36 | 38
  Sudden worsen mood, Week 6/EW, NS | 1 | 0
  Sudden worsen mood, Week 6/EW, OS but worse | 6 | 8
  Sudden worsen mood, Week 6/EW, OS but improved | 9 | 13
  Sudden worse mood, Week 6/EW, OS; unchanged/absent | 53 | 45
  Sudden worsen mood, 7-D FU, NS | 1 | 0
  Sudden worsen mood, 7-D FU, OS but worse | 6 | 6
  Sudden worsen mood, 7-D FU, OS but improved | 11 | 8
  Sudden worsen mood, 7-D FU, OS unchanged/absent | 47 | 48
  Sudden worsened mood, 28-D FU, NS | 3 | 0
  Sudden worsened mood, 28-D FU, OS but worse | 9 | 4
  Sudden worsened mood, 28-D FU, OS but improved | 5 | 8
  Sudden worsed mood, 28-D FU, OS; unchanged/absent | 41 | 47
  Sudden anger outburst, Week 6/EW, NS | 1 | 1
  Sudden anger outburst, Week 6/EW, OS but worse | 5 | 5
  Sudden anger outburst, Week 6/EW, OS but improved | 8 | 9
  Sudden anger outburst,Week 6EW,OS unchanged/absent | 55 | 51
  Sudden anger outburst, 7-D FU, NS | 2 | 1
  Sudden anger outburst, 7-D FU, OS but worse | 4 | 5
  Sudden anger outburst, 7-D FU, OS but improved | 7 | 8
  Sudden anger outburst,7-D FU, OS unchanged/absent | 52 | 48
  Sudden anger outburst, 28-D FU, NS | 1 | 0
  Sudden anger outburst, 28-D FU, OS but worse | 4 | 2
  Sudden anger outburst, 28-D FU, OS but improved | 7 | 7
  Sudden anger outburst, 28-D FU, OS unchang/absent | 45 | 50
  Sudden anger outburst, 28-D FU,missing | 1 | 0
  Sudden panic/anxiety, Week 6/EW, NS | 1 | 0
  Sudden panic/anxiety, Week 6/EW, OS but worse | 5 | 3
  Sudden panic/anxiety, Week 6/EW, OS but improved | 4 | 10
  Sudden panic/anxiety, Wk 6/EW, OS;unchanged/absent | 59 | 53
  Sudden panic/anxiety, 7-D FU, NS | 2 | 0
  Sudden panic/anxiety , 7-D FU, OS but worse | 3 | 1
  Sudden panic/anxiety , 7-D FU, OS but improved | 3 | 7
  Sudden panic/anxiety, 7-D FU, OS unchange/absent | 57 | 54
  Sudden panic/anxiety, 28-D FU, NS | 2 | 0
  Sudden panic/anxiety, 28-D FU, OS; worse | 5 | 1
  Sudden panic/anxiety, 28-D FU, OS; improved | 5 | 8
  Sudden panic/anxiety, 28-D FU,OS; unchanged/absent | 46 | 50
  Bouts of cry/tear, Week 6/EW, NS | 0 | 1
  Bouts of cry/tear, Week 6/EW, OS but worse | 9 | 7
  Bouts of cry/tear, Week 6/EW, OS but improved | 16 | 12
  Bouts of cry/tear, Week 6/EW, OS unchanged/absent | 44 | 46
  Bouts of cry/tear, 7-D FU, NS | 1 | 0
  Bouts of cry/tear, 7-D FU, OS but worse | 8 | 7
  Bouts of cry/tear, 7-D FU, OS but improved | 6 | 11
  Bouts of cry/tear, 7-D FU, OS unchanged/absent | 50 | 44
  Bouts of cry/tear, 28-D FU, NS | 1 | 2
  Bouts of cry/tear, 28-D FU, OS but worse | 8 | 7
  Bouts of cry/tear, 28-D FU, OS but improved | 11 | 10
  Bouts of cry/tear, 28-D FU, OS unchanged/absent | 37 | 40
  Bouts of cry/tear, 28-D FU, missing | 1 | 0
  Agitation, Week 6/EW, NS | 1 | 2
  Agitation, Week 6/EW, OS but worse | 6 | 5
  Agitation, Week 6/EW, OS but improved | 8 | 13
  Agitation, Week 6/EW, OS but unchanged/absent | 54 | 46
  Agitation, 7-D FU, NS | 3 | 0
  Agitation, 7-D FU, OS but worse | 5 | 5
  Agitation, 7-D FU, OS but improved | 5 | 10
  Agitation, 7-D FU, OS but unchanged/absent | 52 | 47
  Agitation, 28-D FU, OS but worse | 6 | 5
  Agitation, 28-D FU, OS but improved | 5 | 6
  Agitation, 28-D FU, OS but unchanged/absent | 46 | 48
  Agitation, 28-D FU, missing | 1 | 0
  Unreal/detached feel, Week 6, NS | 4 | 2
  Unreal/detached feel, Week 6, OS but worse | 4 | 1
  Unreal/detached feel, Week 6, OS but improved | 7 | 7
  Unreal/detached feel, Week 6, OS unchanged/absent | 54 | 56
  Unreal/detached feel, 7-D FU, NS | 2 | 1
  Unreal/detached feel, 7-D FU, OS but worse | 4 | 2
  Unreal/detached feel, 7-D FU, OS but improved | 5 | 5
  Unreal/detached feel, 7-D FU, OS unchanged/absent | 54 | 54
  Unreal/detached feel, 28-D FU, NS | 1 | 1
  Unreal/detached feel, 28-D FU, OS but worse | 4 | 2
  Unreal/detached feel, 28-D FU, OS but improved | 4 | 7
  Unreal/detached feel, 28-D FU, OS;unchanged/absent | 48 | 49
  Unreal/detached feel, 28-D FU, missing | 1 | 0
  Confusion, Week 6/EW, NS | 1 | 0
  Confusion, Week 6/EW, OS but worse | 10 | 8
  Confusion, Week 6/EW, OS but improved | 11 | 15
  Confusion, Week 6/EW, OS but unchanged/absent | 47 | 43
  Confusion, 7-D FU, NS | 1 | 0
  Confusion, 7-D FU, OS but worse | 3 | 7
  Confusion, 7-D FU, OS but improved | 14 | 11
  Confusion, 7-D FU, OS but unchanged/absent | 47 | 44
  Confusion, 28-D FU, NS | 1 | 2
  Confusion, 28-D FU, OS but worse | 7 | 3
  Confusion, 28-D FU, OS but improved | 10 | 12
  Confusion, 28-D FU, OS but unchanged/absent | 40 | 42
  Forgetfulness, Week 6/EW, NS | 1 | 0
  Forgetfulness, Week 6/EW, OS but worse | 9 | 9
  Forgetfulness, Week 6/EW, OS but improved | 8 | 12
  Forgetfulness, Week 6/EW, OS but unchanged/absent | 51 | 45
  Forgetfulness, 7-D FU, NS | 1 | 0
  Forgetfulness, 7-D FU, OS but worse | 4 | 7
  Forgetfulness, 7-D FU, OS but improved | 8 | 7
  Forgetfulness, 7-D FU, OS but unchanged/absent | 52 | 48
  Forgetfulness, 28-D FU, NS | 0 | 1
  Forgetfulness, 28-D FU, OS but worse | 6 | 8
  Forgetfulness, 28-D FU, OS but improved | 7 | 9
  Forgetfulness, 28-D FU, OS but unchanged/absent | 45 | 41
  Mood swings, Week 6/EW, NS | 2 | 0
  Mood swings, Week 6/EW, OS but worse | 7 | 7
  Mood swings, Week 6/EW, OS but improved | 11 | 8
  Mood swings, Week 6/EW, OS but unchanged/absent | 49 | 51
  Mood swings, 7-D FU, NS | 1 | 0
  Mood swings, 7-D FU, OS but worse | 7 | 7
  Mood swings, 7-D FU, OS but improved | 10 | 9
  Mood swings, 7-D FU, OS but unchanged/absent | 47 | 46
  Mood swings, 28-D FU, NS | 1 | 1
  Mood swings, 28-D FU, OS but worse | 9 | 3
  Mood swings, 28-D FU, OS but improved | 6 | 8
  Mood swings, 28-D FU, OS but unchanged/absent | 42 | 47
  Insomnia, Week 6/EW, OS but worse | 7 | 10
  Insomnia, Week 6/EW, OS but improved | 15 | 18
  Insomnia, Week 6/EW, OS but unchanged/absent | 47 | 38
  Insomnia, 7-D FU, NS | 1 | 1
  Insomnia, 7-D FU, OS but worse | 2 | 7
  Insomnia, 7-D FU, OS but improved | 17 | 13
  Insomnia, 7-D FU, OS but unchanged/absent | 45 | 41
  Insomnia, 28-D FU, OS but worse | 13 | 7
  Insomnia, 28-D FU, OS but improved | 10 | 13
  Insomnia, 28-D FU, OS but unchanged/absent | 35 | 39
  Increased dreams, Week 6/EW, NS | 2 | 4
  Increased dreams, Week 6/EW, OS but worse | 2 | 3
  Increased dreams, Week 6/EW, OS but improved | 3 | 6
  Increased dreams, Week 6/EW, OS unchanged/absent | 62 | 53
  Increased dreams, 7-D FU, NS | 3 | 2
  Increased dreams, 7-D FU, OS but worse | 0 | 2
  Increased dreams, 7-D FU, OS but improved | 5 | 4
  Increased dreams, 7-D FU, OS unchanged/absent | 57 | 54
  Increased dreams, 28-D FU, NS | 2 | 3
  Increased dreams, 28-D FU, OS but worse | 3 | 2
  Increased dreams, 28-D FU, OS but improved | 5 | 8
  Increased dreams, 28-D FU, OS unchanged/absent | 48 | 46
  More sweating, Week 6/EW, NS | 1 | 1
  More sweating, Week 6/EW, OS but worse | 1 | 5
  More sweating, Week 6/EW, OS but improved | 3 | 3
  More sweating, Week 6/EW, OS but unchanged/absent | 64 | 57
  More sweating, 7-D FU, NS | 3 | 1
  More sweating, 7-D FU, OS but worse | 1 | 6
  More sweating, 7-D FU, OS but improved | 2 | 6
  More sweating, 7-D FU, OS but unchanged/absent | 59 | 49
  More sweating, 28-D FU, NS | 1 | 2
  More sweating, 28-D FU, OS but worse | 0 | 3
  More sweating, 28-D FU, OS but improved | 4 | 5
  More sweating, 28-D FU, OS but unchanged/absent | 52 | 49
  More sweating, 28-D FU, missing | 1 | 0
  Shake/tremble, Week 6/EW, NS | 1 | 0
  Shake/tremble, Week 6/EW, OS but worse | 2 | 0
  Shake/tremble, Week 6/EW, OS but improved | 6 | 5
  Shake/tremble, Week 6/EW, OS but unchanged/absent | 60 | 61
  Shake/tremble, 7-D FU, NS | 2 | 0
  Shake/tremble, 7-D FU, OS but worse | 3 | 1
  Shake/tremble, 7-D FU, OS but improved | 2 | 3
  Shake/tremble, 7-D FU, OS but unchanged/absent | 58 | 58
  Shake/tremble, 28-D FU, NS | 1 | 1
  Shake/tremble, 28-D FU, OS but worse | 1 | 0
  Shake/tremble, 28-D FU, OS but improved | 2 | 5
  Shake/tremble, 28-D FU, OS but unchanged/absent | 53 | 53
  Shake/tremble, Missing | 1 | 0
  Muscle tension, Week 6/EW, NS | 2 | 1
  Muscle tension, Week 6/EW, OS but worse | 4 | 5
  Muscle tension, Week 6/EW, OS but improved | 8 | 10
  Muscle tension, Week 6/EW, OS but unchanged/absent | 55 | 50
  Muscle tension, 7-D FU, NS | 1 | 1
  Muscle tension, 7-D FU, OS but worse | 3 | 2
  Muscle tension, 7-D FU, OS but improved | 4 | 8
  Muscle tension, 7-D FU, OS but unchanged/absent | 57 | 51
  Muscle tension, 28-D FU, NS | 1 | 0
  Muscle tension, 28-D FU, OS but worse | 3 | 2
  Muscle tension, 28-D FU, OS but improved | 1 | 6
  Muscle tension, 28-D FU, OS but unchanged/absent | 52 | 51
  Muscle ache, Week 6/EW, NS | 1 | 0
  Muscle ache, Week 6/EW, OS but worse | 6 | 5
  Muscle ache, Week 6/EW, OS but improved | 7 | 12
  Muscle ache, Week 6/EW, OS but unchanged/absent | 55 | 49
  Muscle ache, 7-D FU, NS | 1 | 0
  Muscle ache, 7-D FU, OS but worse | 3 | 5
  Muscle ache, 7-D FU, OS but improved | 5 | 9
  Muscle ache, 7-D FU, OS but unchanged/absent | 56 | 48
  Muscle ache, 28-D FU, NS | 2 | 1
  Muscle ache, 28-D FU, OS but worse | 4 | 1
  Muscle ache, 28-D FU, OS but improved | 3 | 6
  Muscle ache, 28-D FU, OS but unchanged/absent | 48 | 51
  Muscle ache, 28-D FU, missing | 1 | 0
  Restless leg, Week 6/EW, NS | 0 | 0
  Restless leg, Week 6/EW, OS but worse | 4 | 4
  Restless leg, Week 6/EW, OS but improved | 4 | 5
  Restless leg, Week 6/EW, OS but unchanged/absent | 61 | 57
  Restless leg, 7-D FU, NS | 0 | 0
  Restless leg, 7-D FU, OS but worse | 3 | 1
  Restless leg, 7-D FU, OS but improved | 2 | 5
  Restless leg, 7-D FU, OS but unchanged/absent | 60 | 56
  Restless leg, 28-D FU, NS | 2 | 1
  Restless leg, 28-D FU, OS but worse | 5 | 1
  Restless leg, 28-D FU, OS but improved | 3 | 4
  Restless leg, 28-D FU, OS but unchanged/absent | 48 | 53
  Muscle cramps, Week 6/EW, NS | 1 | 0
  Muscle cramps, Week 6/EW, OS but worse | 3 | 2
  Muscle cramps, Week 6/EW, OS but improved | 3 | 7
  Muscle cramps, Week 6/EW, OS but unchanged/absent | 62 | 57
  Muscle cramps, 7-D FU, NS | 2 | 2
  Muscle cramps, 7-D FU, OS but worse | 3 | 3
  Muscle cramps, 7-D FU, OS but improved | 3 | 9
  Muscle cramps, 7-D FU, OS but unchanged/absent | 57 | 48
  Muscle cramps, 28-D FU, OS but worse | 3 | 1
  Muscle cramps, 28-D FU, OS but improved | 1 | 5
  Muscle cramps, 28-D FU, OS but unchanged/absent | 53 | 53
  Muscle cramps, 28-D FU, missing | 1 | 0
  Fatigue, Week 6/EW, NS | 1 | 0
  Fatigue, Week 6/EW, OS but worse | 10 | 8
  Fatigue, Week 6/EW, OS but improved | 15 | 17
  Fatigue, Week 6/EW, OS but unchanged/absent | 43 | 41
  Fatigue, 7-D FU, NS | 2 | 1
  Fatigue, 7-D FU, OS but worse | 8 | 9
  Fatigue, 7-D FU, OS but improved | 10 | 9
  Fatigue, 7-D FU, OS but unchanged/absent | 45 | 43
  Fatigue, 28-D FU, NS | 2 | 2
  Fatigue, 28-D FU, OS but worse | 7 | 5
  Fatigue, 28-D FU, OS but improved | 8 | 7
  Fatigue, 28-D FU, OS but unchanged/absent | 41 | 45
  Incoordination, Week 6/EW, NS | 0 | 1
  Incoordination, Week 6/EW, OS but worse | 3 | 1
  Incoordination, Week 6/EW, OS but improved | 2 | 4
  Incoordination, Week 6/EW, OS but unchanged/absent | 64 | 60
  Incoordination, 7-D FU, NS | 1 | 1
  Incoordination, 7-D FU, OS but worse | 0 | 2
  Incoordination, 7-D FU, OS but improved | 1 | 4
  Incoordination, 7-D FU, OS but unchanged/absent | 63 | 55
  Incoordination, 28-D FU, OS but worse | 2 | 2
  Incoordination, 28-D FU, OS but improved | 3 | 3
  Incoordination, 28-D FU, OS but unchanged/absent | 52 | 54
  Incoordination, 28-D FU, missing | 1 | 0
  Blurred vision, Week 6/EW, NS | 2 | 1
  Blurred vision, Week 6/EW, OS but worse | 2 | 0
  Blurred vision, Week 6/EW, OS but improved | 1 | 3
  Blurred vision, Week 6/EW, OS but unchanged/absent | 64 | 62
  Blurred vision, 7-D FU, NS | 1 | 1
  Blurred vision, 7-D FU, OS but improved | 2 | 4
  Blurred vision, 7-D FU, OS but unchanged/absent | 62 | 57
  Blurred vision, 28-D FU, NS | 1 | 0
  Blurred vision, 28-D FU, OS but worse | 3 | 1
  Blurred vision, 28-D FU, OS but improved | 0 | 2
  Blurred vision, 28-D FU, OS but unchanged/absent | 53 | 56
  Blurred vision, 28-D FU, missing | 1 | 0
  Sore eyes, Week 6/EW, NS | 1 | 2
  Sore eyes, Week 6/EW, OS but worse | 1 | 1
  Sore eyes, Week 6/EW, OS but improved | 0 | 3
  Sore eyes, Week 6/EW, OS but unchanged/absent | 67 | 60
  Sore eyes, 7-D FU, NS | 1 | 1
  Sore eyes, 7-D FU, OS but worse | 0 | 1
  Sore eyes, 7-D FU, OS but improved | 2 | 4
  Sore eyes, 28-D FU, NS | 0 | 2
  Sore eyes, 7-D FU, OS but unchanged/absent | 62 | 56
  Sore eyes, 28-D FU, OS but worse | 2 | 1
  Sore eyes, 28-D FU, OS but improved | 0 | 3
  Sore eyes, 28-D FU, OS but unchanged/absent | 55 | 53
  Sore eyes, Missing | 1 | 0
  Uncontrol mouth move, Week 6/EW, NS | 2 | 2
  Uncontrol mouth move, Week 6/EW, OS but improved | 0 | 3
  Uncontrol mouth move,Week6/EW,OS unchanged/absent | 67 | 61
  Uncontrol mouth move, 7-D FU, NS | 1 | 1
  Uncontrol mouth move, 7-D FU, OS but worse | 0 | 1
  Uncontrol mouth move, 7-D FU, OS but improved | 1 | 3
  Uncontrol mouth move, 7-D FU,OS unchanged/absent | 63 | 57
  Uncontrol mouth move, 28-D FU, NS | 0 | 1
  Uncontrol mouth move, 28-D FU, OS but worse | 2 | 1
  Uncontrol mouth move, 28-D FU, OS but improved | 2 | 5
  Uncontrol mouth move,28-D FU, OS unchanged/absent | 53 | 52
  Uncontrol mouth move, missing | 1 | 0
  Speech problem, Week 6/EW, NS | 0 | 1
  Speech problem, Week 6/EW, OS but worse | 1 | 1
  Speech problem, Week 6/EW, OS but improved | 4 | 4
  Speech problem, Week 6/EW, OS but unchanged/absent | 64 | 60
  Speech problem, 7-D FU, OS but worse | 0 | 3
  Speech problem, 7-D FU, OS but improved | 4 | 3
  Speech problem, 7-D FU, OS but unchanged/absent | 61 | 56
  Speech problem, 28-D FU, NS | 1 | 0
  Speech problem, 28-D FU, OS but improved | 3 | 5
  Speech problem, 28-D FU, OS but unchanged/absent | 53 | 54
  Speech problem, 28-D FU, missing | 1 | 0
  Headache, Week 6/EW, NS | 4 | 2
  Headache, Week 6/EW, OS but worse | 5 | 4
  Headache, Week 6/EW, OS but improved | 12 | 10
  Headache, Week 6/EW, OS but unchanged/absent | 48 | 50
  Headache, 7-D FU, NS | 2 | 1
  Headache, 7-D FU, OS but worse | 4 | 3
  Headache, 7-D FU, OS but improved | 12 | 6
  Headache, 7-D FU, OS but unchanged/absent | 47 | 52
  Headache, 28-D FU, NS | 1 | 3
  Headache, 28-D FU, OS but worse | 5 | 2
  Headache, 28-D FU, OS but improved | 6 | 7
  Headache, 28-D FU, OS but unchanged/absent | 46 | 47
  Increased saliva, Week 6/EW, NS | 0 | 0
  Increased saliva, Week 6/EW, OS but worse | 2 | 0
  Increased saliva, Week 6/EW, OS but improved | 0 | 2
  Increased saliva, Week 6/EW, OS unchanged/absent | 67 | 64
  Increased saliva, 7-D FU, NS | 0 | 1
  Increased saliva, 7-D FU, OS but improved | 3 | 2
  Increased saliva, 7-D FU, OS unchanged/absent | 62 | 59
  Increased saliva, 28-D FU, OS but improved | 3 | 3
  Increased saliva, 28-D FU, OS unchanged/absent | 54 | 56
  Increased saliva, 28-D FU, missing | 1 | 0
  Dizziness, Week 6/EW, NS | 2 | 5
  Dizziness, Week 6/EW, OS but worse | 3 | 1
  Dizziness, Week 6/EW, OS but improved | 3 | 2
  Dizziness, Week 6/EW, OS but unchanged/absent | 61 | 58
  Dizziness, 7-D FU, NS | 3 | 1
  Dizziness, 7-D FU, OS but worse | 3 | 1
  Dizziness, 7-D FU, OS but improved | 4 | 4
  Dizziness, 7-D FU, OS but unchanged/absent | 55 | 56
  Dizziness, 28-D FU, OS but worse | 4 | 1
  Dizziness, 28-D FU, NS | 0 | 0
  Dizziness, 28-D FU, OS but improved | 1 | 3
  Dizziness, 28-D FU, OS but unchanged/absent | 53 | 55
  Nose running, Week 6/EW, NS | 2 | 2
  Nose running, Week 6/EW, OS but worse | 0 | 1
  Nose running, Week 6/EW, OS but improved | 5 | 3
  Nose running, Week 6/EW, OS but unchanged/absent | 62 | 60
  Nose running, 7-D FU, NS | 1 | 3
  Nose running, 7-D FU, OS but improved | 3 | 2
  Nose running, 7-D FU, OS but unchanged/absent | 61 | 57
  Nose running, 28-D FU, NS | 0 | 1
  Nose running, 28-D FU, OS but worse | 1 | 0
  Nose running, 28-D FU, OS but improved | 1 | 3
  Nose running, 28-D FU, OS but unchanged/absent | 55 | 55
  Nose running, 28-D FU, missing | 1 | 0
  Breath shortness, Week 6/EW, NS | 0 | 1
  Breath shortness, Week 6/EW, OS but improved | 3 | 2
  Breath shortness, Week 6/EW, OS unchanged/absent | 66 | 63
  Breath shortness, 7-D FU, NS | 0 | 1
  Breath shortness, 7-D FU, OS but improved | 3 | 4
  Breath shortness, 7-D FU, OS unchanged/absent | 62 | 57
  Breath shortness, 28-D FU, OS but worse | 0 | 2
  Breath shortness, 28-D FU, OS but improved | 1 | 2
  Breath shortness, 28-D FU, OS unchanged/absent | 56 | 55
  Breath shortness, 28-D FU, missing | 1 | 0
  Chills, Week 6/EW, NS | 1 | 1
  Chills, Week 6/EW, OS but worse | 0 | 1
  Chills, Week 6/EW, OS but improved | 4 | 2
  Chills, Week 6/EW, OS but unchanged/absent | 64 | 62
  Chills, 7-D FU, NS | 1 | 1
  Chills, 7-D FU, OS but worse | 1 | 2
  Chills, 7-D FU, OS but improved | 1 | 2
  Chills, 7-D FU, OS but unchanged/absent | 62 | 57
  Chills, 28-D FU, NS | 0 | 1
  Chills, 28-D FU, OS but worse | 1 | 0
  Chills, 28-D FU, OS but improved | 1 | 4
  Chills, 28-D FU, OS but unchanged/absent | 55 | 54
  Chills, 28-D FU, missing | 1 | 0
  Fever, Week 6/EW, OS but improved | 2 | 1
  Fever, Week 6/EW, OS but unchanged/absent | 67 | 65
  Fever, 7-D FU, NS | 0 | 1
  Fever, 7-D FU, OS but improved | 2 | 2
  Fever, 7-D FU, OS but unchanged/absent | 63 | 59
  Fever, 28-D FU, OS but improved | 0 | 3
  Fever, 28-D FU, OS but unchanged/absent | 57 | 56
  Fever, 28-D FU, missing | 1 | 0
  Vomiting, Week 6/EW, OS but worse | 0 | 1
  Vomiting, Week 6/EW, OS but improved | 3 | 1
  Vomiting, Week 6/EW, OS but unchanged/absent | 66 | 64
  Vomiting, 7-D FU, NS | 1 | 1
  Vomiting, 7-D FU, OS but improved | 2 | 3
  Vomiting, 7-D FU, OS but unchanged/absent | 62 | 58
  Vomiting, 28-D FU, OS but worse | 1 | 0
  Vomiting, 28-D FU, OS but improved | 1 | 2
  Vomiting, 28-D FU, OS but unchanged/absent | 56 | 57
  Nausea, Week 6/EW, NS | 2 | 0
  Nausea, Week 6/EW, OS but worse | 4 | 2
  Nausea, Week 6/EW, OS but improved | 4 | 2
  Nausea, Week 6/EW, OS but unchanged/absent | 59 | 62
  Nausea, 7-D FU, NS | 5 | 1
  Nausea, 7-D FU, OS but worse | 1 | 2
  Nausea, 7-D FU, OS but improved | 4 | 4
  Nausea, 7-D FU, OS but unchanged/absent | 55 | 55
  Nausea, 28-D FU, NS | 1 | 3
  Nausea, 28-D FU, OS but worse | 3 | 0
  Nausea, 28-D FU, OS but improved | 2 | 4
  Nausea, 28-D FU, OS but unchanged/absent | 52 | 52
  Diarrhea, Week 6/EW, NS | 2 | 0
  Diarrhea, Week 6/EW, OS but worse | 2 | 0
  Diarrhea, Week 6/EW, OS but improved | 2 | 1
  Diarrhea, Week 6/EW, OS but unchanged/absent | 63 | 65
  Diarrhea, 7-D FU, NS | 1 | 1
  Diarrhea, 7-D FU, OS but worse | 0 | 1
  Diarrhea, 7-D FU, OS but improved | 4 | 4
  Diarrhea, 7-D FU, OS but unchanged/absent | 60 | 56
  Diarrhea, 28-D FU, NS | 2 | 1
  Diarrhea, 28-D FU, OS but worse | 0 | 0
  Diarrhea, 28-D FU, OS but improved | 0 | 3
  Diarrhea, 28-D FU, OS but unchanged/absent | 56 | 55
  Stomach cramps, Week 6/EW, NS | 0 | 1
  Stomach cramps, Week 6/EW, OS but worse | 4 | 1
  Stomach cramps, Week 6/EW, OS but improved | 2 | 3
  Stomach cramps, Week 6/EW, OS but unchanged/absent | 63 | 61
  Stomach cramps, 7-D FU, NS | 1 | 1
  Stomach cramps, 7-D FU, OS but worse | 1 | 2
  Stomach cramps, 7-D FU, OS but improved | 4 | 5
  Stomach cramps, 7-D FU, OS but unchanged/absent | 59 | 54
  Stomach cramps, 28-D FU, NS | 0 | 1
  Stomach cramps, 28-D FU, OS but worse | 0 | 1
  Stomach cramps, 28-D FU, OS but improved | 3 | 2
  Stomach cramps, 28-D FU, OS but unchanged/absent | 55 | 55
  Stomach bloat, Week 6/EW, NS | 1 | 3
  Stomach bloat, Week 6/EW, OS but worse | 4 | 2
  Stomach bloat, Week 6/EW, OS but improved | 1 | 5
  Stomach bloat, Week 6/EW, OS but unchanged/absent | 63 | 56
  Stomach bloat, 7-D FU, NS | 2 | 2
  Stomach bloat, 7-D FU, OS but worse | 1 | 0
  Stomach bloat, 7-D FU, OS but improved | 3 | 5
  Stomach bloat, 7-D FU, OS but unchanged/absent | 59 | 55
  Stomach bloat, 28-D FU, NS | 0 | 2
  Stomach bloat, 28-D FU, OS but worse | 0 | 1
  Stomach bloat, 28-D FU, OS but improved | 3 | 4
  Stomach bloat, 28-D FU, OS but unchanged/absent | 54 | 52
  Stomach bloat, 28-D FU, Missing | 1 | 0
  Unusual vision, Week 6/EW, NS | 2 | 1
  Unusual vision, Week 6/EW, OS but worse | 1 | 1
  Unusual vision, Week 6/EW, OS but improved | 1 | 3
  Unusual vision, Week 6/EW, OS but unchanged/absent | 65 | 61
  Unusual vision, 7-D FU, NS | 1 | 0
  Unusual vision, 7-D FU, OS but improved | 2 | 3
  Unusual vision, 7-D FU, OS but unchanged/absent | 62 | 59
  Unusual vision, 28-D FU, OS but worse | 1 | 1
  Unusual vision, 28-D FU, OS but improved | 1 | 3
  Unusual vision, 28-D FU, OS but unchanged/absent | 55 | 55
  Unusual vision, 28-D FU, missing | 1 | 0
  Sense of burn, Week 6/EW, NS | 1 | 1
  Sense of burn, Week 6/EW, OS but worse | 1 | 0
  Sense of burn, Week 6/EW, OS but improved | 1 | 2
  Sense of burn, Week 6/EW, OS but unchanged/absent | 66 | 63
  Sense of burn, 7-D FU, OS but worse | 0 | 1
  Sense of burn, 7-D FU, OS but improved | 2 | 3
  Sense of burn, 7-D FU, OS but unchanged/absent | 63 | 58
  Sense of burn, 28-D FU, OS but worse | 2 | 0
  Sense of burn, 28-D FU, OS but improved | 1 | 4
  Sense of burn, 28-D FU, OS but unchanged/absent | 54 | 55
  Sense of burn, 28-D FU,missing | 1 | 0
  Unusual sound feel, Week 6/EW, NS | 1 | 1
  Unusual sound feel, Week 6/EW, OS but worse | 3 | 2
  Unusual sound feel, Week 6/EW, OS but improved | 2 | 3
  Unusual sound feel, Week 6/EW, OS unchanged/absent | 63 | 60
  Unusual sound feel, 7-D FU, OS but worse | 1 | 1
  Unusual sound feel, 7-D FU, OS but improved | 3 | 2
  Unusual sound feel, 7-D FU, OS unchanged/absent | 61 | 59
  Unusual sound feel, 28-D FU, OS but worse | 2 | 1
  Unusual sound feel, 28-D FU, OS but improved | 1 | 4
  Unusual sound feel, 28-D FU, OS unchanged/absent | 54 | 54
  Unusual sound feel, 28-D FU, missing | 1 | 0
  Noise in ear, Week 6/EW, NS | 0 | 1
  Noise in ear, Week 6/EW, OS but worse | 1 | 0
  Noise in ear, Week 6/EW, OS but improved | 1 | 4
  Noise in ear, Week 6/EW, OS but unchanged/absent | 67 | 61
  Noise in ear, 7-D FU, OS but worse | 0 | 1
  Noise in ear, 7-D FU, OS but improved | 2 | 2
  Noise in ear, 7-D FU, OS but unchanged/absent | 63 | 59
  Noise in ear, 28-D FU, OS but worse | 1 | 0
  Noise in ear, 28-D FU, OS but improved | 1 | 4
  Noise in ear, 28-D FU, missing | 1 | 0
  Noise in ear, 28-D FU, OS but unchanged/absent | 55 | 55
  Unusual taste/smell, Week 6/EW, OS but worse | 1 | 0
  Unusual taste/smell, Week 6/EW, OS but improved | 2 | 2
  Unusual taste/smell, Week 6/EW,OS unchanged/absent | 66 | 64
  Unusual taste/smell, 7-D FU, NS | 1 | 0
  Unusual taste/smell, 7-D FU, OS but worse | 0 | 1
  Unusual taste/smell, 7-D FU, OS but improved | 2 | 3
  Unusual taste/smell, 7-D FU, OS unchanged/absent | 62 | 58
  Unusual taste/smell, 28-D FU, OS but improved | 1 | 2
  Unusual taste/smell, 28-D FU, OS unchanged/absent | 56 | 57
  Unusual taste/smell, 28-D FU, missing | 1 | 0

ADVERSE EVENTS:
Time Frame: Up to 28 Day Follow-up (18 months)
Description: All Subject Population
Arm/Group | GSK561679 | Placebo
All-Cause Mortality (participants affected / at risk) | 0/74 | 0/76
Serious Adverse Events (participants affected / at risk) | 0/74 | 1/76
Other Adverse Events (participants affected / at risk) | 34/74 | 44/76
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | GSK561679 (N=74) | Placebo (N=76)
Breast cancer stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GSK561679 (N=74) | Placebo (N=76)
Headache (Nervous system disorders) | 9 (9) | 17 (19)
Nausea (Gastrointestinal disorders) | 15 (18) | 10 (10)
Nasopharyngitis (Infections and infestations) | 6 (6) | 5 (5)
Dry mouth (Gastrointestinal disorders) | 5 (5) | 5 (5)
Diarrhoea (Gastrointestinal disorders) | 3 (3) | 5 (5)
Constipation (Gastrointestinal disorders) | 5 (5) | 2 (2)
Dizziness (Nervous system disorders) | 3 (3) | 4 (4)
Fatigue (General disorders) | 2 (2) | 5 (5)
Vomiting (Gastrointestinal disorders) | 2 (3) | 4 (4)
Flatulence (Gastrointestinal disorders) | 1 (1) | 4 (4)
Insomnia (Psychiatric disorders) | 4 (4) | 1 (1)
Irritability (General disorders) | 0 (0) | 4 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.